CLINICAL TRIAL: NCT04856397
Title: Ozurdex in Suboptimal Diabetic Macular Edema
Brief Title: Ozurdex in Suboptimal Diabetic Macular Edema Patients
Acronym: DME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Principal Investigator, Sohel Somani, Principal Investigator, Uptown Eye Specialists
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2020-06-29; First posted 2021-04-23 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Calcium Dobesilate; aflibercept

STUDY DESIGN:
Intervention Model Description: There are four cohorts of patients in this study (please see below on study procedures). To be able to have meaningful data showing statistical significance, we will need at least 30 patients in each cohort of patients, accounting for There will be at least 30 patients in each cohort. We will need at least 100 patients enrolled in the study prior to randomization of the non-responders into early switch (~30) or late switch (~30) or non-switch (~30). The estimated number also accounts for the estimated number of patients who will be lost to follow-up or may drop out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Other): Responders will be in this category. These patients will be maintained on intravitreal anti-VEGF therapy for 1 year, with a monthly PRN ("as needed") treatment regimen post 5 monthly loading doses.
  Interventions: Drug: Eylea
- Early switch (Experimental): Suboptimal responders who are switched to intravitreal Ozurdex (monitored monthly and treated PRN at a potential 2-6 month interval) injections after the first 3 monthly loading intravitreal eylea.
  Interventions: Drug: Intravitreal Implant in Applicator; Drug: Eylea
- Late switch (Experimental): Suboptimal responders who are switched to intravitreal Ozurdex (monitored monthly and treated PRN at a potential 2-6 month interval) injections after the first 6 monthly loading intravitreal eylea
  Interventions: Drug: Intravitreal Implant in Applicator; Drug: Eylea
- Non-switch (Other): Suboptimal responders who continue to receive monthly intravitreal anti-VEGF injections.
  Interventions: Drug: Eylea

INTERVENTIONS:
Drug: Intravitreal Implant in Applicator — Dexamethasone intravitreal implant
  Other Names: Ozurdex
  Arms: Early switch; Late switch
Drug: Eylea — anti-VEGF medication

SUMMARY:
The primary focus of this study is to understand the anatomic and visual outcomes of patients with refractory and suboptimal treatment response diabetic macular edema (DME) using anti-vascular endothelial growth factor (VEGF) to Ozurdex, an intravitreal dexamethasone implant. Secondly, investigators aim to understand the differences in cytokine profiles in patients who respond differently to intravitreal anti-VEGF versus Ozurdex. The importance of this study is to identify biomarkers that may help predict patients' response to different treatment protocols. Currently, Ozurdex is not covered by provincial health benefit plans for patients with DME. Our results may help improve access to care for those who have suboptimal results with or refractory to intravitreal anti-VEGF treatment.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) is the most common cause of vision loss in young patients with diabetes. Its pathophysiology starts with decreased retinal oxygen tension that manifests as retinal capillary hyperpermeability and increased intravascular pressure mediated by vascular endothelial growth factor (VEGF) upregulation and retinal vascular autoregulation, respectively. Spectral domain optical coherence tomography (SD-OCT) is the cornerstone of clinical assessment of DME. The foundation of treatment is metabolic control of hyperglycemia and blood pressure. Specific ophthalmic treatments of DME include intravitreal anti-VEGF drug injections, in the form of intravitreal Bevacizumab (Avastin), Ranibizumab (Lucentis), and Aflibercept (Eylea). Intravitreal corticosteroid injections, focal laser photocoagulation, and vitrectomy are other treatment options. A substantial fraction of eyes respond incompletely to all of these modalities resulting in visual loss and disordered retinal structure and vasculature visible on SD-OCT and OCT angiography. There is currently no consensus on when to switch from one treatment to another in the context of a suboptimal response. Our hypothesis is that patients who are switched early to Ozurdex and achieve an OCT proven dry state, achieve better functional outcomes than those patients who are switched late or not at all, by limiting exposure of the retina to potentially damaging inflammatory markers, and the merits associated with less frequent injections.

Suboptimal DME is defined as a central subfoveal retinal thickness of > 300 and the presence of intra or sub-retinal fluid with a minimum BCVA of 20/25 or worse after 3 injections of intravitreal aflibercept, from here on referred to as Eylea. Furthermore, there is some evidence that a subset of patients with refractory DME respond well to intravitreal corticosteroids, specifically, Ozurdex, which is a biodegradable, sustained-release intravitreal dexamethasone implant, designed to be potentially injected between 2-6 months. This medication is currently not covered by the Ontario health benefits plan for patients with DME and comes at a significant cost to patients.

Moreover, recent studies have confirmed the important role of inflammatory ocular cytokines in patients' response to intravitreal treatments in DME, much the same as neovascular age-related macular degeneration. However, it is not known which ocular cytokines determine the degree of response to various treatment modalities for DME.

Here, investigators aim to study the anatomic and visual outcomes, as well as the cytokine profile of patients with suboptimal DME in response to early vs. late switch to intravitreal Ozurdex treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-native patients with DME secondary to type I or type II diabetes mellitus
2. Patients who require intravitreal anti-VEGF treatment
3. Able to understand English and complete a pain assessment
4. Suboptimal DME responders in patients who have received 3 or 6 eylea injections (non-cytokine group)

Exclusion Criteria:

1. Deafness or communication disorder, known Dementia, Severe COPD/Asthma (severe lung disorder), Severe OSA, Psychiatric or Anxiety conditions, involuntary movement disorders, allergy to the anesthesia, any conditions requiring intraoperative iris manipulation, any prior ocular surgery; all patients who may need translation, are illiterate, or unable to provide consent.
2. Pre-existing ocular pathology confounding outcome (i.e. uveitis, retinal vascular disease, macular degeneration etc.)
3. Pre-existing uncontrolled glaucoma/high IOP
4. Patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-25 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  best corrected visual acuity (BCVA)

SECONDARY OUTCOMES:
OCT findings | 1 year
  Track anatomic outcomes on optical coherence tomography (OCT)
OCTa findings | 1 year
  Track anatomic outcomes on optical coherence tomography angiography (OCTA)
Cytokine expression TNFa | 1 year
  baseline cytokine profile of the aqueous humour of all patients prior to first dose of anti-VEGF. Cytokine TNFa
Cytokine expression IL-8 | 1 year
  baseline cytokine profile of the aqueous humour of all patients prior to first dose of anti-VEGF. Cytokine IL-8
Cytokine expression IL-6 | 1 year
  baseline cytokine profile of the aqueous humour of all patients prior to first dose of anti-VEGF. Cytokine IL-6

IPD SHARING:
Plan to Share IPD: No